CLINICAL TRIAL: NCT03260660
Title: Comparison of MR Elastography Methods Without and With Compressed Sensing
Status: Completed | Type: Observational
Sponsor: Children's Hospital Medical Center, Cincinnati (Other)
Responsible Party: Sponsor
Other Study IDs: CIN_CompMRE_001
Record Dates: First submitted 2017-08-14; First posted 2017-08-24 (Actual); Last update posted 2018-01-29 (Actual); Status verified 2018-01

CONDITIONS: Liver Diseases
MeSH Terms: conditions — Liver Diseases | interventions — Elasticity Imaging Techniques

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

INTERVENTIONS:
Device: Magnetic Resonance Elastography — The investigators plan to prospectively assess the agreement of liver stiffness measurements obtained using standard of care MR elastography techniques vs. MR elastography with varying amounts of imaging acceleration using compressed sensing in adult volunteers

SUMMARY:
In this research study, the investigators will compare the liver stiffness results obtained from the current Magnetic Resonance Imaging (MRI) method to liver stiffness results obtained from a method that uses faster imaging techniques.

DETAILED DESCRIPTION:
MR elastography is increasingly used to assess liver stiffness in pediatric and adult patients with chronic liver diseases. While numerous tissue abnormalities can affect liver stiffness, liver stiffness measured by MR elastography is most often used to predict and quantify liver fibrosis. Conventional MR elastography techniques require multiple breath-holds that are 12-20 seconds in length. In the pediatric population, reliable breath-holding >10 seconds can be challenging. Recently, compressed sensing has become available as a method for accelerating image data acquisition, and thus shortening breath-holds.

ELIGIBILITY:
Inclusion Criteria:

* Adult volunteers ≥18 years of age
* Ability to tolerate 30 minutes in an MRI scanner.
* Nothing to eat or drink for 4 hours prior to the MRI scan

Exclusion Criteria:

* No contraindication to MR imaging (e.g., implanted non-MRI compatible device)
* Known or suspected pregnancy. Female subjects of child bearing potential will undergo a urine pregnancy test prior to imaging.

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Healthy Volunteers
Sampling Method: Non-Probability Sample
Enrollment: 25 (Actual)
Dates: Start 2017-08-15 (Actual); Primary Completion 2017-12-01 (Actual); Study Completion 2017-12-01 (Actual)

PRIMARY OUTCOMES:
Standard Magnetic Resonance Elastography versus Elastography with Compressed Sensing (x1.5) | 30 minutes
  Four MR elastography images through the mid liver will be obtained using standard MR elastography and MR elastography with 1.5 times the amount of standard Sensing applied. Correlation Coefficient will be determined for resulting elastography data.
Standard Magnetic Resonance Elastography versus Elastography with Compressed Sensing (x2) | 30 minutes
  Four MR elastography images through the mid liver will be obtained using standard MR elastography and MR elastography with 2 times the amount of standard sensing applied. correlation coefficient will be determined for resulting elastography data.
Standard Magnetic Resonance Elastography versus Elastography with Compressed Sensing (x3) | 30 minutes
  Four MR elastography images through the mid liver will be obtained using standard MR elastography and MR elastography with 3 times the amount of standard Sensing applied. Correlation coefficient will be determined for resulting elastography data.

SECONDARY OUTCOMES:
Standard Magnetic Resonance Elastography versus respiratory triggered Magnetic Resonance Elastography. | 30 minutes
  Four MR elastography images through the mid liver will be obtained using standard MR elastography and MR elastography acquired using respiratory triggered Gradient Recalled Elastography. Correlation coefficient will be determined for resulting elastography data.
Standard Magnetic Resonance Elastography versus navigated triggered Magnetic Resonance Elastography. | 30 minutes
  Four MR elastography images through the mid liver will be obtained using standard MR elastography and MR elastography acquired using navigated triggered Gradient Recalled Elastography. Correlation coefficient will be determined for resulting elastography data.

CONTACTS AND LOCATIONS:
Overall Officials: Jonathan Dillman, MD,MSc, Principal Investigator — Children's Hospital Medical Center, Cincinnati
Locations (1):
- Cincinnati Children's Hospital Medical Center, Cincinnati, Ohio, United States

IPD SHARING:
Plan to Share IPD: No